CLINICAL TRIAL: NCT01733862
Title: A Study to Assess the Impact of Rotavirus Vaccination on Hospitalizations and Outpatient Visits Due to Rotavirus Gastroenteritis (RV GE) in Japan
Brief Title: Study to Assess the Impact of Vaccination on Hospitalizations and Outpatient Visits Due to Rotavirus Gastroenteritis
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116929
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Infections, Rotavirus; Rotavirus Vaccines
Keywords: Impact; Vaccination; Hospitalizations; Rotavirus gastroenteritis; Japan
MeSH Terms: conditions — Rotavirus Infections; Tooth, Impacted | interventions — Data Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Group Japan: Children less than five years of age, hospitalized for RV GE or AGE and children with outpatient or emergency room visits for RV GE or AGE, between November 2007 and October 2016 (i.e., before and after the introduction of RV vaccination in Japan) in any of the selected hospitals.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data sheet. Data will be collected and is planned to be analysed at the following time points:
  Pre-vaccination period: Nov 2007 to Oct 2011, transition period: Nov 2011 to Oct 2012 and post vaccination period: Nov 2012 to Oct 2016.

SUMMARY:
This study aims at assessing the impact of RV vaccination in hospitals in Nagoya City (administrative district), Japan, where RV vaccines have been introduced since November 2011 and financial support for vaccination costs by Nagoya city, Japan have been implemented from October 2012.

DETAILED DESCRIPTION:
The electronic admission database or any other applicable database of the hospital will be reviewed to identify hospitalized children/children with outpatient visits/emergency room visits, less than five years of age who had been diagnosed with acute gastroenteritis (AGE) or RV GE either by the International Classification of Diseases and Related Health Problems 10th Revision (ICD 10) diagnostic code (AA00-AA09 for intestinal infectious diseases and A08.0 for RV specific GE) or by RV positive rapid diagnosis kit results.

Note: The outcomes for the outpatient and emergency room visits will be assessed only in case the data for outpatient and emergency room visits can be obtained from at least one of the study centers.

ELIGIBILITY:
Inclusion Criteria:

- Children aged less than five years visiting hospitals for RV GE or AGE from 2007 to 2016, who live in the study area.

Exclusion Criteria:

- Not applicable.

Max Age: 1824 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include children less than five years of age, hospitalized for RV GE or AGE and children with outpatient or emergency room visits for RV GE or AGE, between November 2007 and October 2016 (i.e., before and after the introduction of RV vaccination in Japan) in any of the selected hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 5394 (Actual)
Dates: Start 2012-11-27 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of RV GE hospitalizations among all hospitalized children aged less than five years. | From Nov 2007 to Oct 2016

SECONDARY OUTCOMES:
Occurrence of RV GE hospitalizations among AGE hospitalizations in children less than five years of age. | From Nov 2007 to Oct 2016
Occurrence of RV GE hospitalizations by age group in children less than five years of age. | From Nov 2007 to Oct 2016
Occurrence of AGE hospitalizations among all hospitalized children aged less than five years. | From Nov 2007 to Oct 2016
Occurrence of outpatient visits for AGE among all outpatient visits in children less than five years of age. | From Nov 2007 to Oct 2016
Occurrence of outpatient visits for RV GE among all outpatient visits in children less than five years of age. | From Nov 2007 to Oct 2016
Occurrence of outpatient visits for RV GE among AGE outpatient visits in children less than five years of age. | From Nov 2007 to Oct 2016
Duration of hospitalizations for RV GE or AGE, overall, for each year, season in children less than five years of age. | From Nov 2007 to Oct 2016
Occurrence of hospitalizations for RV GE among all emergency visits for RV GE in children less than five years of age. | From Nov 2007 to Oct 2016

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Aichi, Japan

REFERENCES:
- [Background] Yoshikawa T, Matsuki T, Sato K, Mizuno M, Shibata M, Hasegawa S, Morita M, Iwasa M, Gopala K, Holl K. Impact of rotavirus vaccination on the burden of acute gastroenteritis in Nagoya city, Japan. Vaccine. 2018 Jan 25;36(4):527-534. doi: 10.1016/j.vaccine.2017.12.006. Epub 2017 Dec 13. PMID 29248263
- See also: Results Summary, Full Protocol and Analysis Plan for study 116929 can be found on the GSK Clinical Study Register — https://www.gsk-studyregister.com/study/4892